CLINICAL TRIAL: NCT04952181
Title: Optical Biometry Versus Ultrasonic Biometry in Intraocular Lens Calculation in High Myopic Cataractous Patients: A Comparative Study
Brief Title: Comparison Between Different Investigations Used in Intraocular Lens Calculation in High Myopic Cataractous Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Ahmed Okasha, principle investigator, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-21-06-01
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Calculation of Intraocular Lens in High Myopic Cataractous Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optical biometry (Experimental)
  Interventions: Device: optical biometry
- ultrasonic biometry (Experimental)
  Interventions: Device: ultrasonic biometry

INTERVENTIONS:
Device: optical biometry — optical biometry is a fast, noncontact method it uses the method of partial coherence interferometry (PCI) to measure the axial length (AXL), based on reflection of the interference signal of the retinal pigment epithelium.
  Arms: optical biometry
Device: ultrasonic biometry — ultrasonic biometry is contact method depends on ultrasonic transducer producing thin sound beam travelling through different media of the eye when it faces interface of substance dissimilar from that it is travelling through part is reflecting and the other travel through the different substance
  Arms: ultrasonic biometry

SUMMARY:
the purpose of the study is to compare the accuracy of optical and ultrasonic biometry in intraocular lens (IOL) calculation in high myopic cataractous patients

DETAILED DESCRIPTION:
* Prospective interventional (QUASI experimental) comparative study
* This study will be conducted on high myopic cataractous patients scheduled for phacoemulsification and IOL implantation in department of ophthalmology, Sohag university
* patients will be divided into 2 groups one will be subjected to intraocular lens (IOL) calculation by optical biometry the second one will be subjected to intraocular lens (IOL) calculation by ultrasonic biometry
* postoperative auto refraction after I month

ELIGIBILITY:
Inclusion Criteria:

* patients with simple cataract not associated with other pathologies suitable for phacoemulsification and 1ry IOL implantation With axial length (AXL) equal to or greater than 26.5mm

Exclusion Criteria:

1. History of trauma
2. Associated pathologies such as optic neuropathy, age related macular degeneration, macular edema, retinal detachment, , ocular inflammation, retinitis pigmentosa, proliferative diabetic retinopathy
3. corneal opacities or irregularities, scars, dystrophy or ectasia
4. Patients who underwent previous corneal surgery (including refractive surgery)
5. Patients having intraoperative complications as inability to achieve secure 'in the bag' placement of the IOL (i.e. due to posterior capsule rupture, vitreous loss, weak zonules, or zonular rupture)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
desired post operative refraction | postoperative refraction 1 month
  detection of postoperative refraction by the use of autorefractor (one of the objective methods of assessment of refraction) after use of IOL power calculated by different investigations (optical vs ultrasonic)

REFERENCES:
- [Background] Tappeiner C, Rohrer K, Frueh BE, Waelti R, Goldblum D. Clinical comparison of biometry using the non-contact optical low coherence reflectometer (Lenstar LS 900) and contact ultrasound biometer (Tomey AL-3000) in cataract eyes. Br J Ophthalmol. 2010 May;94(5):666-7. doi: 10.1136/bjo.2009.167700. No abstract available. PMID 20447976
- [Background] Wang L, Shirayama M, Ma XJ, Kohnen T, Koch DD. Optimizing intraocular lens power calculations in eyes with axial lengths above 25.0 mm. J Cataract Refract Surg. 2011 Nov;37(11):2018-27. doi: 10.1016/j.jcrs.2011.05.042. PMID 22018365
- [Background] Olsen T. Improved accuracy of intraocular lens power calculation with the Zeiss IOLMaster. Acta Ophthalmol Scand. 2007 Feb;85(1):84-7. doi: 10.1111/j.1600-0420.2006.00774.x. PMID 17244216